CLINICAL TRIAL: NCT05984030
Title: Meet me Where I am: A Multilevel Strategy to Increase PrEP Uptake and Persistence in Rural NC
Brief Title: Supporting Tailored And Responsive PrEP in Rural North Carolina
Acronym: STARR-NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-3058; R61AI174285 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: HIV Pre-Exposure Prophylaxis

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to Intervention Condition or Control Condition. The study will use blocked randomization stratified by county, with randomly ordered blocks of sizes 4 and 6.
  Depending on their date of enrollment, participants will be asked to complete baseline and quarterly assessments at 3, 6, and 12-month follow-ups. Primary outcome measures are assessed at month 3. Secondary outcome measures are assessed at months 3 and 6.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STARR NC Intervention Condition (Experimental): Intervention arm will receive a multilevel intervention with three components: a PrEP Navigator to facilitate linkage to PrEP services and completion of applications for health insurance/drug assistance; a Digital Health Intervention (DHI) platform (HealthMpowerment); and referral to Telehealth PrEP services as an option for linking to PrEP care.
  The Intervention Arm version of the DHI includes: Study Timeline and Calendar, publicly-available PrEP locator feature, Dried Blood Spot self-collection kit ordering, Educational Health Resource Center; Interactive skill-building health activities; social support newsfeed/group chat; Ask the Expert anonymous health question and answer; Medication Tracker; Health Behavior Tracker; Gamification features for participant engagement.
  Intervention Arm participants will complete baseline and quarterly follow-up assessments.
  Intervention Arm participants will complete two Dried Blood Spot self-collection kits at 3 and 6 months.
  Interventions: Other: PrEP Navigation Services; Other: Telehealth PrEP Services Referral; Behavioral: HealthMpowerment Digital Health Intervention - Enhanced
- STARR NC Standard-of-Care Control Condition (Active Comparator): Standard-of-Care Control arm will receive the standard PrEP referral services available at the STI clinic setting where they were recruited. They will also receive study staff guided support to install the control arm version of the HealthMPowerment DHI platform.
  The Control Arm version of the DHI includes: Study Timeline and Calendar, publicly-available PrEP locator feature, Dried Blood Spot self-collection kit ordering, Educational Health Resource Center.
  Control Arm participants will complete baseline and quarterly follow-up assessments.
  Control Arm participants will complete two Dried Blood Spot self-collection kits at 3 and 6 months.
  Interventions: Behavioral: HealthMpowerment Digital Health Intervention - Basic

INTERVENTIONS:
Other: PrEP Navigation Services — Trained professional PrEP navigators will connect with intervention arm participants following study onboarding. Primary navigator responsibilities include helping participants engage in PrEP care, assisting with completing necessary paperwork for insurance, referral to PrEP care, and application for drug assistance programs, as needed. Navigation services will be available to participants for the first 6 months of participation (active intervention period). Navigation services are tailored to the individual needs of each intervention arm participant
  Arms: STARR NC Intervention Condition
Other: Telehealth PrEP Services Referral — PrEP Navigators can link interested intervention arm participants to telehealth PrEP services via self-referral. The study facilitates referral for intervention arm participants to pre-existing telehealth PrEP services. The telehealth PrEP services participants receive are not provided, financed, or staffed by the study. Participants will receive telehealth PrEP services via the technology platform or service that the provider typically employs. PrEP clinical eligibility, visit frequency, monitoring labs, and all other PrEP management will be at the discretion of the established PrEP provider. PrEP navigators can assist with appointment scheduling, reminders, and other provider-access issues, as requested, for the first 6 months of study participation.
  Arms: STARR NC Intervention Condition
Behavioral: HealthMpowerment Digital Health Intervention - Enhanced — The Enhanced version of the HealthMpowerment Digital Health Intervention includes all features from the Basic version, plus the following additional features: Interactive skill-building health activities; social support newsfeed/group chat; Ask the Expert anonymous health question and answer; Medication Tracker; Health Behavior Tracker; Gamification features for participant engagement.
  Arms: STARR NC Intervention Condition
Behavioral: HealthMpowerment Digital Health Intervention - Basic — The Control Arm version of the HealthMpowerment Digital Health Intervention includes: Study Timeline and Calendar, publicly-available PrEP locator feature, Dried Blood Spot self-collection kit ordering, Educational Health Resource Center.
  Arms: STARR NC Standard-of-Care Control Condition

SUMMARY:
This project consists of two phases to be completed over five years. Phase 1 (Aims 1 and 2) will be completed during Years 1-3 (R61). The Phase 1 study is a randomized trial of a multilevel HIV Pre-Exposure Prophylaxis (PrEP) intervention strategy in rural and peri-urban North Carolina sexually transmitted infection (STI) clinics, with primary outcome of PrEP uptake within 3 months of an index STI clinic visit.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to an intervention or control condition. Participants enrolled in the intervention arm will receive a multilevel intervention with three components: a PrEP Navigator to facilitate linkage to PrEP services and completion of applications for health insurance/drug assistance; a Digital Health Intervention (DHI) platform (HealthMpowerment) - a HIPAA-compliant evidence-based DHI that provides interactive educational resources, social support, and tools for developing PrEP behavioral skills and self-efficacy; and referral to Telehealth PrEP services as an option for linking to PrEP care.

Control arm participants will receive the standard PrEP referral services available at the STI clinic setting where they were recruited. They will also receive linkage to a limited version of the DHI, with basic PrEP resources and information.

ELIGIBILITY:
Inclusion Criteria:

* Report sexual activity with a male in the past 12 months
* Received HIV testing within 90 days pre-enrollment and not known to be HIV-positive at screening/enrollment by self-report
* Age 18-39 years
* Have daily smartphone access
* Be English speaking
* Deny current PrEP use

Exclusion Criteria:

* Confirmed prior HIV-positive diagnosis
* Prior PrEP use (oral PrEP or injectable PrEP) within the last 3 months.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants assigned female at birth must identify as cisgender to be eligible for participation.
Enrollment: 17 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rutstein, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following publication of primary study results.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Rutstein SE, Ferguson E, Mansour O, Brown N, Stocks JB, Washington A, Mobley V, Dowler S, Edwards J, Hightow-Weidman LB, Hurt CB, Pence B, Muessig KE. Multilevel Intervention to Support Tailored and Responsive HIV Pre-Exposure Prophylaxis Care in Rural North Carolina: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 21;14:e68085. doi: 10.2196/68085. PMID 40117579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prospective participants deemed study-eligible are required to complete the following before being randomized and enrolled in the study: (1) informational video, (2) informed consent, (3) HIPAA authorization, (4) baseline survey. To continue study participation, participants must receive baseline HIV testing and be confirmed seronegative within 45 days of completing the pre-screening questionnaire. Participants who do not verify HIV-negative status within that 45-day window are study-stopped.
Groups:
- STARR NC Intervention Condition: Intervention arm will receive a multilevel intervention with three components: a PrEP Navigator; an enhanced version of the Digital Health Intervention (DHI) platform (HealthMpowerment); and referral to Telehealth PrEP services as an option for linking to PrEP care.
  Intervention Arm participants will complete baseline and quarterly follow-up assessments, and two Dried Blood Spot self-collection kits at 3 and 6 months.
  PrEP Navigation Services: Primary navigator responsibilities include helping participants engage in PrEP care, assisting with completing necessary paperwork for insurance, referral to PrEP care, and application for drug assistance programs. Navigation services will be available to participants for the first 6 months of participation.
  Telehealth PrEP Services Referral: PrEP Navigators can link intervention arm participants to pre-existing telehealth PrEP services via self-referral. PrEP navigators can assist with appointment scheduling, reminders, and other provider-access issues, as requested, for the first 6 months of study participation.
  HealthMpowerment Digital Health Intervention - Enhanced: The Enhanced version includes all features from the Basic version, plus the following: Interactive skill-building health activities; social support newsfeed/group chat; Ask the Expert anonymous health question and answer; Medication Tracker; Health Behavior Tracker.
- STARR NC Standard-of-Care Control Condition: Standard-of-Care Control arm will receive the standard PrEP referral services available at the STI clinic setting where they were recruited. They will also receive study staff guided support to install the control arm version of the HealthMPowerment DHI platform.
  The Control Arm version of the DHI includes: Study Timeline and Calendar, publicly-available PrEP locator feature, Dried Blood Spot self-collection kit ordering, Educational Health Resource Center.
  Control Arm participants will complete baseline and quarterly follow-up assessments.
  Control Arm participants will complete two Dried Blood Spot self-collection kits at 3 and 6 months.
  HealthMpowerment Digital Health Intervention - Basic: The Control Arm version of the HealthMpowerment Digital Health Intervention includes: Study Timeline and Calendar, publicly-available PrEP locator feature, Dried Blood Spot self-collection kit ordering, Educational Health Resource Center.
Period: Overall Study
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Started | 7 | 10
Completed | 6 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 1 | 4 | 5
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Reporting PrEP Initiation by 3 Months
Description: Proportion of participants with verified self-reported pre-exposure prophylaxis (PrEP) use (first dose, oral or injectable PrEP)1 at or before 3 months, defined as the number verified to start PrEP divided by the total number of participants in each arm
Time Frame: 3 months
Measure: Number; unit: proportion of participants
Groups:
- STARR NC Intervention Condition: Intervention arm will receive a multilevel intervention with three components: a PrEP Navigator; an enhanced version of the Digital Health Intervention (DHI) platform (HealthMpowerment); and referral to Telehealth PrEP services as an option for linking to PrEP care.
- STARR NC Standard-of-Care Control Condition: Standard-of-Care Control arm will receive the standard PrEP referral services available at the STI clinic setting where they were recruited. They will also receive study staff guided support to install the control arm version of the HealthMPowerment DHI platform.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 6 | 10
proportion of participants | 0.33 | 0.10

2. Secondary Outcome: Proportion of Participants Reporting PrEP Initiation by 6 Months
Description: Proportion of participants with verified self-reported PrEP use (first dose, oral or injectable PrEP) at or before 6 months, defined as the number verified to start PrEP divided by the total number of participants in each arm
Time Frame: 6 months
Population: Of the 16 participants enrolled who were followed through study completion, 12 participants were enrolled before 10/01/2024 and eligible for 6 months of follow-up.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 4 | 8
proportion of participants | 0.50 | 0.13

3. Secondary Outcome: Proportion of PrEP Initiators Adhering to Chosen PrEP Strategy Over First 3 Months
Description: Number of participants with on-time PrEP refills and/or injections noted in Electronic Health Record (EHR) over first 3 months divided by number initiating PrEP over first 3 months
Time Frame: 3 months
Population: All available data are reported. Of the 16 participants enrolled who were followed through study completion, only 3 participants initiated PrEP over the first 3 months. The 2 intervention PrEP initiators had available PrEP refill data, while the 1 control participant PrEP initiator did not.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
proportion of participants | 0.50 | 0.00

4. Secondary Outcome: Proportion of PrEP Initiators Adhering to Chosen PrEP Strategy Over First 6 Months
Description: Number of participants with on-time PrEP refills and/or injections noted in EHR over first 6 months divided by number initiating PrEP over first 6 months
Time Frame: 6 months
Population: All available data are collected. Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, only 3 initiated PrEP in the first 6 months. One of the two intervention participants had available PrEP refill data. The control participant PrEP initiator did not have available PrEP refill data.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
proportion of participants | 0.00 | 0.00

5. Secondary Outcome: Average Number of Consecutive Months PrEP Used Over First 3 Months
Description: Among those who initiate PrEP, average number of consecutive months PrEP used, based on date of first and last dose over first 3 months of follow-up, as indicated through survey self-report and visits/prescriptions noted in the EHR.
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, only 3 participants initiated PrEP in the first 3 months.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
months | 1.76 (0.21) | 3.29 (NA) — No standard deviation can be calculated as only one participant is contributing data for this metric.

6. Secondary Outcome: Average Number of Consecutive Months PrEP Used Over First 6 Months
Description: Among those who initiate PrEP, average number of consecutive months PrEP used, based on date of first and last dose over first 6 months of follow-up, as indicated through survey self-report and visits/prescriptions noted in the EHR
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, only 3 participants initiated PrEP.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
months | 1.34 (0.79) | 3.29 (NA) — No standard deviation can be calculated as only one participant is contributing data for this metric.

7. Secondary Outcome: Average Number of Days PrEP Used Among Persons Initiating Daily Oral PrEP in the 30 Days Prior to the 3-month Visit.
Description: Among those who initiate daily oral PrEP, average number of days PrEP used, based on self-reported recall of doses taken in past 30 days.
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, only 3 participants initiated PrEP over the first 3 months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
days | 16.50 (16.26) | 28.00 (NA) — No standard deviation can be calculated as only one participant is contributing data for this metric

8. Secondary Outcome: Average Number of Condomless Anal Sex Acts Protected by PrEP Among Persons Initiating Event-driven Oral PrEP in the 30 Days Prior to the 3-month Visit.
Description: Among those who initiate event-driven oral PrEP, average number of condomless anal sex acts covered by PrEP, based on self-reported number of condomless anal sex episodes and frequency of complete event-driven PrEP use (before and after) condomless anal sex act.
Time Frame: 3-months
Population: Of the 16 participants enrolled who were followed through study completion, none of the participants initiated event-driven oral PrEP.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Proportion of Injectable PrEP Initiators Reporting PrEP Use in the 90 Days Prior to the 3-month Visit
Description: Number of participants who initiated injectable PrEP and reported using Injectable PrEP within an on-time injection interval, in the 90 days prior to the 3-month visit, divided by the number who initiated injectable PrEP.
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, none of the participants initiated injectable PrEP.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Average Number of Days PrEP Used Among Persons Initiating Daily Oral PrEP in the 30 Days Prior to the 6-month Visit.
Description: as for outcome 7
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, 3 participants initiated PrEP, but only 2 of those participants initiated PrEP before the 6-month visit.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 1 | 1
Days | 0 (NA) — No standard deviation can be calculated as only one participant is contributing data for this metric. | 0 (NA) — No standard deviation can be calculated as only one participant is contributing data for this metric.

11. Secondary Outcome: Average Number of Condomless Anal Sex Acts Protected by PrEP Among Persons Initiating Event-driven Oral PrEP in the 30 Days Prior to the 6-month Visit.
Description: Among those who initiate event-driven oral PrEP, average proportion of condomless anal sex acts covered by PrEP, based on self-reported number of condomless anal sex episodes and frequency of complete event-driven PrEP use (before and after) condomless anal sex act.
Time Frame: 6 months
Population: Of the 12 participants enrolled who were enrolled before 10/01/2024 and followed for 6 months, none of the participants initiated event-driven oral PrEP.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Proportion of Injectable PrEP Initiators Reporting PrEP Use in the 90 Days Prior to the 6-month Visit
Description: as for outcome 9
Time Frame: 6 months
Population: Of the 12 participants enrolled who were enrolled before 10/01/2024 and followed for 6 months, none of the participants initiated injectable PrEP.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Proportion of Oral PrEP Initiators With Detected PrEP Concentrations in Blood at 3 Months
Description: Number of PrEP initiators with PrEP concentrations detected at the 3-month study follow-up visit, based on intraerythrocytic Tenofovir diphosphate (TFV-DP) collected as Dried Blood Spot (DBS) divided by the number who initiated oral PrEP
Time Frame: 3 months
Population: as for outcome 7
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
proportion of participants | 0.00 | 0.00

14. Secondary Outcome: Proportion of Oral PrEP Initiators With Detected PrEP Concentrations in Blood at 6 Months
Description: Number of PrEP initiators with PrEP concentrations detected at the 6-month study follow-up visit, based on intraerythrocytic TFV-DP collected as DBS divided by the number who initiated oral PrEP
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, only 3 participants initiated PrEP in the first 6 months.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 1
proportion of participants | 0.00 | 0.00

15. Secondary Outcome: Proportion of Injectable PrEP Initiators Receiving All Prescribed Injections Through 3 Months
Description: Number of injectable PrEP initiators with injections recorded in the EHR at all prescribed timepoints prior to the 3-month follow up visit divided by the number who initiated injectable PrEP
Time Frame: 3 months
Population: as for outcome 9
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Proportion of Injectable PrEP Initiators Receiving All Prescribed Injections Through 6 Months
Description: Number of injectable PrEP initiators with injections recorded in the EHR at all prescribed timepoints prior to the 6-month follow up visit divided by the number who initiated injectable PrEP
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, none of the participants initiated injectable PrEP.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Proportion of Participants Who Test Positive for HIV Among Those Tested at or Prior to the 3-month Visit
Description: Number with a positive clinical test result for human immunodeficiency virus (HIV) obtained from state, clinic, or commercial lab results, or verified participant-uploaded results, divided by the number tested for HIV prior to the 3-month visit, as indicated by state, clinic, commercial, or self-uploaded indication of receiving a test
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, only 2 participants received HIV testing at or prior to the 3-month visit.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 0
proportion of participants | 0.00 |

18. Secondary Outcome: Proportion of Participants Who Test Positive for HIV Among Those Tested at or Prior to the 6-month Visit
Description: Number with a positive clinical test result for HIV obtained from state, clinic, or commercial lab results, or verified participant-uploaded results, divided by the number tested for HIV prior to the 6-month visit, as indicated by state, clinic, commercial, or self-uploaded indication of receiving a test
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, only 2 participants received HIV testing at or prior to the 6-month visit.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 0
proportion of participants | 0.00 |

19. Secondary Outcome: Proportion of Participants Who Test Positive for an STI Other Than HIV Among Those Tested at or Prior to the 3-month Visit
Description: Number with a positive clinical test result for an sexually transmitted infections (STI) other than HIV obtained from state, clinic, or commercial lab results, or verified participant-uploaded results, divided by the number tested for STIs other than HIV prior to the 3 month visit, as indicated by state, clinic, commercial, or self-uploaded indication of receiving a test
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, only 2 participants received STI testing at or prior to the 3-month visit.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 0
proportion of participants | 0.00 |

20. Secondary Outcome: Proportion of Participants Who Test Positive for an STI Other Than HIV Among Those Tested at or Prior to the 6-month Visit
Description: Number with a positive clinical test result for an STI other than HIV obtained from state, clinic, or commercial lab results, or verified participant-uploaded results, divided by the number tested for STIs other than HIV prior to the 6-month visit, as indicated by state, clinic, commercial, or self-uploaded indication of receiving a test.
Time Frame: 6 months
Population: Of the 12 participants who enrolled before 10/01/2024 and were eligible for 6 months of follow-up, only 2 participants received STI testing at or prior to the 6-month visit.
Measure: Number; unit: proportion of participants
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 2 | 0
proportion of participants | 0.00 |

21. Secondary Outcome: Average Self-reported Score on the PrEP Stigma Scale at 3 Months
Description: Average self-reported score on the PrEP Anticipated Stigma Scale as reported on the computer-assisted self-interview (CASI) at 3 months
  The mean composite score is calculated from the PrEP Anticipated Stigma Scale (Calabrese et al., 2018), an 8-item validated scale measuring the sub-constructs of PrEP user stereotypes and PrEP disapproval by others. Item response options include: (1) Strongly Disagree, (2) Disagree, (3) Agree, (4) Strongly Agree. Mean scores are calculated, with higher scores indicating stronger perceived PrEP stigma. Total possible composite score ranges from 8 (lowest stigma, best outcome) to 32 (highest stigma, worst outcome).
Time Frame: 3 months
Population: Of the 16 participants enrolled who were followed through study completion, only 12 participants responded to the 3M PrEP Anticipated Stigma survey questions.
Measure: Mean (Standard Deviation); unit: score on PrEP Stigma Scale
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 5 | 7
score on PrEP Stigma Scale | 15.80 (3.35) | 16.71 (3.15)

22. Secondary Outcome: Average Self-reported Score on the PrEP Stigma Scale at 6 Months
Description: Average self-reported score on the PrEP Anticipated Stigma Scale as reported on the CASI at 6 months
  The mean composite score is calculated from the PrEP Anticipated Stigma Scale (Calabrese et al., 2018), an 8-item validated scale measuring the sub-constructs of PrEP user stereotypes and PrEP disapproval by others. Item response options include: (1) Strongly Disagree, (2) Disagree, (3) Agree, (4) Strongly Agree. Mean scores are calculated, with higher scores indicating stronger perceived PrEP stigma. Total possible composite score ranges from 8 (lowest stigma, best outcome) to 32 (highest stigma, worst outcome).
Time Frame: 6 months
Population: Of the 12 participants enrolled before 10/01/2024 and eligible for 6 months of follow-up, only 8 participants responded to the 6M PrEP Anticipated Stigma survey questions.
Measure: Mean (Standard Deviation); unit: score on PrEP Stigma Scale
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
Number analyzed (Participants) | 3 | 5
score on PrEP Stigma Scale | 15.33 (1.53) | 14.8 (4.97)

ADVERSE EVENTS:
Time Frame: All participants were followed for a minimum of 3 months. Depending on the date of their study enrollment, participants were followed for 3, 6, or 12 months. Specifically per protocol, participants enrolled before 04/01/2024 were followed for 12 months, participants enrolled before 10/01/2024 were followed for 6 months, and participants enrolled before 01/01/2024 were followed for 3 months.
Arm/Group | STARR NC Intervention Condition | STARR NC Standard-of-Care Control Condition
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT05984030/Prot_SAP_001.pdf
  • Informed Consent Form (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT05984030/ICF_002.pdf